CLINICAL TRIAL: NCT05047653
Title: The Prognostic Value of the Abnormalities on the Chest Radiography Versus the Chest Computed Tomography in Critically Ill COVID-19 Patients - Protocol for a National Study Comparing the RALE With the CORADS and CT-Severity Score
Brief Title: RALE Versus CORADS/CT-Severity Score in COVID-19
Acronym: RALE-CORADS
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Prof. Dr. Marcus J. Schultz, Prof., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: RALE-CORADS
Record Dates: First submitted 2021-09-14; First posted 2021-09-17 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pneumonia
Keywords: RALE score; severity score; CORADS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RALE score vs. severity score — RALE score vs. severity score and CORADS

SUMMARY:
Rationale Patients with severe coronavirus disease 2019 (COVID-19) frequently fulfill the criteria for acute respiratory distress syndrome (ARDS), with extensive and bilateral abnormalities on the chest radiography (CXR) and the chest computed tomography (CT) abnormalities. The 'Radiographic Assessment of Lung Edema' (RALE) score, the 'COVID-19 Reporting and Data System' (CO-RADS) score, and the 'CT severity score' may all have prognostic value in critically ill patients with acute respiratory failure due to COVID-19.

Objectives To compare the prognostic value of the RALE score, the CO-RADS score and the CT severity score in critically ill patients with ARDS due to COVID-19.

Hypotheses The RALE score, the CO-RADS score and the CT severity score have prognostic value (primary). The RALE score, the CO-RADS score and the CT severity score correlate well.

Study design National, retrospective observational study. Study population Critically ill COVID-19 patients with acute respiratory failure, who received at least one CXR and one chest CT scan during critical illness.

Method CXRs are visually scored by two independent investigators, using the RALE score approach. Chest CT scans are scored by an independent radiologist, using the CO-RADS score and the CT severity score. Demographic, ventilation and outcome data are captured from the hospital systems.

Main study parameters/endpoints ICU mortality (primary) and hospital-, 28-, 90-mortality, the number of days alive and free from invasive ventilation, duration of ventilation in survivors, and length of stay in ICU and hospital.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Participants will not directly benefit from participation, but burden is absent. The CRX and chest CT scans have already been obtained as part of routine clinical care. Collecting CXR for RALE scoring and chest CT scans for CO-RADS and CT severity scoring, clinical and outcome data is of no harm for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* admitted to the intensive care unit of the Amsterdam UMC, location 'AMC', between March 1, 2020 and May 31, 2020 (the first 3 months of the first wave of the national outbreak in the Netherlands) and between October 1, 2020 and December 31, 2020 (the first 3 months of the second wave in the Netherlands);
* RT-PCR confirmed coronavirus diseases 2019 (COVID-19); and
* having had received at least one chest radiograph (CXR) and one adjacent chest computed tomography (CT) scan during the period a patient was having acute respiratory failure.

Exclusion Criteria:

* Age < 18 years.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Invasive ventilated COVID-19 patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
ICU mortality | 90 days
  The ICU mortality with a maximum of 90 days

SECONDARY OUTCOMES:
hospital mortality | 90 days
  The hospital mortality with a maximum of 90 days
28-day mortality | 28 days
  The 28-day mortality
90-day mortality | 90 days
  The 90-day mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA), Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided